CLINICAL TRIAL: NCT01636466
Title: Zortress (Everolimus) to Prevent Alloantibody Formation in Patients With Late Stage Renal Allograft Failure: The Everolimus-Transplant Exit Strategy Trial (E-TEST)
Brief Title: The Everolimus-Transplant Exit Strategy Trial (E-TEST)
Acronym: E-TEST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Feasibility
Sponsor: Ashtar Chami (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Ashtar Chami, Assistant Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00059278; CRAD001AUS191T (Other: Other)
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Kidney Failure, Chronic
Keywords: Chronic allograft failure; Kidney Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus conversion (Experimental): Subjects who have previously undergone a kidney transplant and are in late stage renal allograft failure will be randomized to take everolimus 0.75 mg twice daily after discontinuing current calcineurin inhibitor. Subjects will be weaned off of all other immunosuppression medicines when dialysis starts.
  Interventions: Drug: Everolimus
- Control (No Intervention): Subjects who have previously undergone a kidney transplant and are in late stage renal allograft failure will be randomized to continue on current immunosuppressive regimen. Subjects will be weaned off of all immunosuppression medicines when dialysis starts.

INTERVENTIONS:
Drug: Everolimus — Everolimus will initially be dosed at 0.75 mg tablet taken orally twice a day. The dose will be adjusted to maintain serum trough concentrations of 5-8 ng/ml.
  Other Names: Zortress
  Arms: Everolimus conversion

SUMMARY:
The purpose of this study is to test the safety and effectiveness of everolimus (Zortress®) in preventing antibody formation in patients with chronic failing kidney transplants. Everolimus (Zortress®) is approved by the U.S. Food and Drug Administration for the prevention of rejection in kidney transplant.

The primary objective for the study is to determine whether conversion of patients with chronic renal graft failure approaching dialysis to an everolimus-based regimen will prevent allosensitization. The secondary objective will be to determine whether conversion of patients with chronic renal graft failure to everolimus (elimination of calcineurin inhibitor) will delay the onset of dialysis.

ELIGIBILITY:
Inclusion Criteria:

* recipient of deceased or living donor kidney transplant
* Age 18-75 years (inclusive)
* Male or female
* renal allograft dysfunction/deterioration evidenced by glomerular filtration rate (GFR) less than or equal to 35
* Grade 2 or 3 Interstitial fibrosis/tubular atrophy (IF/TA) on renal allograft biopsy within 5 years of enrollment
* Willing and able to provide informed consent for study participation

Exclusion Criteria:

* Prior solid organ transplant (other than kidney)
* History of donor-specific antibody
* History of biopsy-proven acute rejection within 1 year prior to enrollment
* Proteinuria greater than or equal to 1.5 gm on spot urine protein/creatinine ratio
* Evidence of Hepatitis C virus infection (antibody positive or polymerase chain reaction(PCR) positive)
* Epstein Barr Virus (EBV) or cytomegalovirus (CMV) viremia at the time of enrollment
* Subjects receiving belatacept (Nulojix)
* Pregnant or nursing (lactating) women
* Women of child-bearing potential (WOCBP) who are unwilling or unable to use two birth-control methods throughout participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashtar Chami, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus Conversion: Subjects who have previously undergone a kidney transplant and were in late stage renal allograft failure were randomized to take everolimus at least 0.75 mg twice daily after discontinuing current calcineurin inhibitor. Subjects were weaned off of all other immunosuppression medicines when dialysis started.
- Control: Subjects who have previously undergone a kidney transplant and were in late stage renal allograft failure were randomized to continue on current immunosuppressive regimen. Subjects were weaned off of all immunosuppression medicines when dialysis started.
Period: Overall Study
Arm/Group | Everolimus Conversion | Control
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus Conversion | Control | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Fluorescence Index (MFI) of Donor Specific Alloantibodies (DSA)
Description: Development of new donor-specific alloantibody as determined by solid phase bead array (Luminex) technology defining MFIs for fine specificity at Class I and Class II antigens (human leukocyte antigens (HLA) - A, B, C, DR, DP, and DQ) with an MFI >5000 defined as positive
Time Frame: 36 months
Population: Single subject enrolled was terminated early. Data analysis was not performed as the Month 36 visit did not occur.
Arm/Group | Everolimus Conversion | Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence of Return to Dialysis Dependence
Time Frame: 36 months
Population: Single subject enrolled was terminated early. Data analysis was not performed as the Month 36 visit did not occur.
Arm/Group | Everolimus Conversion | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Everolimus Conversion | Control
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus Conversion (N=1) | Control (N=0)
Pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes